CLINICAL TRIAL: NCT00321880
Title: Healing Touch as a Supportive Intervention for Adult Acute Leukemia Patients: A Pilot Study
Brief Title: Healing Touch in Treating Patients Receiving Chemotherapy for Acute Myeloid Leukemia or Acute Lymphocytic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000471996; CCCWFU-02305; CCCWFU-BG06-006
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2012-07

CONDITIONS: Fatigue; Leukemia; Psychosocial Effects of Cancer and Its Treatment
Keywords: fatigue; psychosocial effects of cancer and its treatment; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia
MeSH Terms: conditions — Fatigue; Leukemia; Congenital Abnormalities; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: therapeutic touch — administration of healing touch in 30 minute sessions

SUMMARY:
RATIONALE: Supportive care, such as healing touch, may improve quality of life in patients receiving chemotherapy for acute leukemia.

PURPOSE: This clinical trial is studying how well healing touch works in treating patients receiving chemotherapy for acute myeloid leukemia or acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of conducting a randomized controlled trial, in terms of recruiting and retaining participants, to a study of healing touch (HT) as supportive care in patients receiving chemotherapy for acute myeloid leukemia or acute lymphoblastic leukemia.
* Examine potential barriers to participation and ascertain reasons for study drop-outs in these patients.
* Demonstrate whether these patients will comply with treatment sessions and remain in the study.
* Obtain preliminary data on the effectiveness of HT on psychological distress and treatment-related symptoms focusing on fatigue and sleep disturbances in these patients.
* Determine if the HT protocol needs to be refined, modified, or eliminated, based on pilot participant feedback, for a randomized clinical trial.

OUTLINE: This is a pilot study.

Within 1 week of admission to the hospital, patients are interviewed by a research assistant about previous use of complementary or alternative medicine therapies, knowledge of healing touch (HT), previous experience with HT, willingness to participate in a study of HT for acute leukemia patients, and willingness to be randomized in a HT study. The first 12 patients interested in undergoing HT undergo a 30-minute session of HT therapy 3 times a week during weeks 2, 3, and 4 of induction or reinduction chemotherapy. Patients are also asked to rate current distress, pain, fatigue, and nausea before and after the second HT session during weeks 2, 3, and 4. Patients also complete self-report questionnaires at baseline, during week 5 of induction or reinduction chemotherapy or prior to discharge from the hospital, and during the first week of consolidation chemotherapy (approximately week 9-13).

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following acute leukemias:

  * Acute lymphocytic leukemia
  * Acute myeloid leukemia
* Hospitalized for induction (newly diagnosed patients) or reinduction (relapsed patients) chemotherapy
* Must be oncology inpatients at Wake Forest University Baptist Medical Center

PATIENT CHARACTERISTICS:

* Must know adequate English to understand the consent form, complete questionnaires, and converse with study staff

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-02; Primary Completion 2007-02 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruiting and retaining patients for a randomized controlled trial to study healing touch (HT) as supportive care | 4 weeks
Effectiveness of healing touch on reducing psychological stress and fatigue | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C. Danhauer, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States